CLINICAL TRIAL: NCT00998426
Title: Evaluation of Blood Glucose Levels for Hepatitis B Immune Globulin (HepaGam B) Administration
Brief Title: Evaluating Blood Glucose Levels During Infusion With HepaGam B (HBIG) in Post-liver Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Cangene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009-337
Record Dates: First submitted 2009-10-07; First posted 2009-10-20 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-04

CONDITIONS: Hepatitis B
Keywords: hepatitis B immune globulin; HBIG; HepaGam B; orthotopic liver transplant
MeSH Terms: conditions — Hepatitis B | interventions — hepatitis B hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All study participants (Experimental): Study procedures will occur one timebetween post-op day 1 and post-op day 7. Study procedures to include blood glucose monitoring prior to and after (various time points for 2 hours after) infusion with HBIG.
  Interventions: Procedure: glucose monitoring before and after HepaGam B administration; Biological: HepaGam B (Hepatitis B Immune Globulin (HBIG))

INTERVENTIONS:
Procedure: glucose monitoring before and after HepaGam B administration — Glucose monitoring before and after HepaGam B administration. Prior to receiving the dose of HepaGam B HBIG, blood glucose will be monitored in 3 manners. These will include two finger stick tests, one with a glucose-specific monitoring device and one with a glucose non-specific monitoring device; a venous blood glucose level; and a urine glucose test. Patients will receive the HBIG infusion and then immediately after the dose will have the same blood glucose tests repeated (finger sticks, venous glucose and urine glucose). Then at 60 minutes and 120 minutes after the dose is given, patients will again have finger stick tests with the glucose specific and glucose non-specific monitoring devices.
  Other Names: HepaGam B; Hepatitis B Immune Globulin
Biological: HepaGam B (Hepatitis B Immune Globulin (HBIG)) — Subjects will be given 20,000 IU HepaGam B after the initial blood glucose monitoring, and prior to the post-infusion blood glucose monitoring.

SUMMARY:
HepaGam B Hepatitis B Immune Globulin (HBIG) solution contains 10% maltose, which could possibly interfere with the measurement of glucose levels when using glucose non-specific tests. The purpose of this study is to determine whether use of HepaGam B HBIG shows an increase in glucose levels in the body using non-specific glucose monitoring, as well as specific glucose monitoring. The sponsor believes that this medication will not cause a significant increase in glucose levels in the body when measured by glucose non-specific tests.

DETAILED DESCRIPTION:
BACKGROUND:

Hepatitis B Immune Globulin (HBIG) is used post liver transplantation (OLT) in hepatitis B surface antigen-positive recipients to prevent recurrence of hepatitis B. One formulation of HBIG, HepaGam B, contains the disaccharide maltose, which can potentially falsely elevate glucose readings when glucose nonspecific point of care (GNSPOC) testing is used, such as a glucose dehydrogenase pyrroloquinolinequinone (GDH-PQQ)-based method. This can result in inappropriate administration of antidiabetic agents and resultant episodes of clinically significant hypoglycemia. Glucose specific point of care (GSPOC) testing, such as a glucose oxidase-based method, however, is not affected by the presence of maltose. The purpose of this study was to determine if there was a significant difference in glucose readings using GSPOC and GNSPOC monitoring devices after HBIG administration.

METHODS:

This is a nonrandomized, prospective study evaluating patients receiving maintenance HBIG therapy over 3 months post liver transplantation. Blood glucose levels in each subject were analyzed by GSPOC and GNSPOC devices at specific times around HBIG administration.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* HBsAG positive candidates for HBV related liver transplant to be placed on HepaGam B therapy for the prevention of HBV recurrence in both the acute phase (immediately post operative) and the long term maintenance phase
* at least 18 years of age

Exclusion Criteria:

* unable or unwilling to provide written informed consent
* concomitant administration of other maltose containing products such as dietary supplements, dietary aids, IVIG, external peritoneal dialysis solution in both arms
* concomitant administration of corticosteroids in the long term maintenance phase
* pregnancy, as determined by a pregnancy test administered after consent has been signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirti Shetty, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult OLT recipients receiving maintenance HBIG therapy were recruited from the inpatient liver transplant service.
Groups:
- All Study Participants: Study procedures will occur one time between post-op day 1 and post-op day 7. These will include blood glucose monitoring prior to and after (various time points for 2 hours after) infusion with HBIG.
  Prior to receiving the dose of HepaGam B HBIG, blood glucose will be monitored in 3 manners. These will include two finger stick tests, one with a glucose-specific monitoring device and one with a glucose non-specific monitoring device; a venous blood glucose level; and a urine glucose test. Patients will receive the HBIG infusion and then immediately after the dose will have the same blood glucose tests repeated (finger sticks, venous glucose and urine glucose). Then at 60 minutes and 120 minutes after the dose is given, patients will again have finger stick tests with the glucose specific and glucose non-specific monitoring devices.Subjects will be given 20,000 IU HepaGam B after the initial blood glucose monitoring, and prior to the post-infusion blood glucose monitoring
Period: Overall Study
Arm/Group | All Study Participants
Started | 5
Blood Glucose Monitoring | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Study procedures will occur one time between post-op day 1 and post-op day 7. These will include blood glucose monitoring prior to and after (various time points for 2 hours after) infusion with HBIG.
  Prior to receiving the dose of HepaGam B HBIG, blood glucose will be monitored in 3 manners. All participants will undergo two finger stick tests, one with a glucose-specific monitoring device(GS-POC) and one with a glucose non-specific monitoring device(GNS-POC) and a venous blood glucose level. Patients will receive the HBIG infusion and then immediately after the dose will have the same blood glucose tests repeated (finger sticks, venous glucose ). Then at 60 minutes and 120 minutes after the dose is given, patients will again have finger stick tests with the glucose specific and glucose non-specific monitoring devices.Subjects will be given 20,000 IU HepaGam B after the initial blood glucose monitoring, and prior to the post-infusion blood glucose monitoring
Arm/Group | All Study Participants
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5
adult OLT recipients [Number; unit: participants] — This is a nonrandomized, prospective study evaluating patients receiving maintenance HBIG therapy over 3 months post liver transplantation. Blood glucose levels in each subject were analyzed by GSPOC and GNSPOC devices at specific times around HBIG administration
  participants | 5

OUTCOME MEASURES:

1. Primary Outcome: Differences in Blood Glucose Levels as Measured by GNS-POC, GS-POC and Venous Blood Prior to and After HBIG Injection
Description: All participants received GNS-POC, GS-POC and venous blood glucose measurements prior to and after HBIG injection( immediately following, 60 and 120 min post dose).
Time Frame: Pre-dose, immediately following, 60 min and 120 min after injection
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- All Study Participants: Study procedures will occur one time between post-op day 1 and post-op day 7. These will include blood glucose monitoring prior to and after (various time points for 2 hours after) infusion with HBIG.
  Prior to receiving the dose of HepaGam B HBIG, blood glucose will be monitored in 3 manners. These will include two finger stick tests, one with a glucose-specific monitoring device (GS-POC)and one with a glucose non-specific (GNS-POC) monitoring device; a venous blood glucose level. Patients will receive the HBIG infusion and then immediately after the dose will have the same blood glucose tests repeated (finger sticks, venous glucose and urine glucose). Then at 60 minutes and 120 minutes after the dose is given, patients will again have finger stick tests with the glucose specific and glucose non-specific monitoring devices.Subjects will be given 20,000 IU HepaGam B after the initial blood glucose monitoring, and prior to the post-infusion blood glucose monitoring
Arm/Group | All Study Participants
Number analyzed (Participants) | 5
mg/dL
  Pre Dose: GNS POC minus GS POC | -3.2 (8.2)
  Post Dose GNS POC minus GS POC | 6.0 (13.5)
  60 minutes GNS POC minus GS POC | 56.6 (125.1)
  120 minutes GNS POC minus GS POC | -2.6 (10.1)
  Predose GNSPOC minus Venous glucose | 7.4 (3.5)
  PredoseGSPOC minus venous blood glucose | 10.6 (6)
  Post-dose GNS POC minus venous blood glucose | 17 (12.5)
  Post-dose GS POC minus venous blood glucose | 11 (25.7)
Statistical Analysis 1: Comparison: All Study Participants; A random intercept model was used to fit the five subjects' glucose reading data over time. The fixed effect glucose meters, time effect and their interactions were included in the model; Test type: Superiority or Other; p = 0.59, Random intercept model — This is the p value for the meter by time interaction

ADVERSE EVENTS:
Groups:
- Acute Phase: Study procedures will occur one time between post-op day 1 and post-op day 7. These will include blood glucose monitoring prior to and after (various time points for 2 hours after) infusion with HBIG.
  Prior to receiving the dose of HepaGam B HBIG, blood glucose will be monitored in 3 manners. These will include two finger stick tests, one with a glucose-specific monitoring device and one with a glucose non-specific monitoring device; a venous blood glucose level; and a urine glucose test. Patients will receive the HBIG infusion and then immediately after the dose will have the same blood glucose tests repeated (finger sticks, venous glucose and urine glucose). Then at 60 minutes and 120 minutes after the dose is given, patients will again have finger stick tests with the glucose specific and glucose non-specific monitoring devices.Subjects will be given 20,000 IU HepaGam B after the initial blood glucose monitoring, and prior to the post-infusion blood glucose monitoring
- Chronic Phase: Study procedures will occur one time at least three (3) months post liver transplant. These will include blood glucose monitoring prior to and after (various time points for 2 hours after) infusion with HBIG.
  glucose monitoring before and after HepaGam B administration: Prior to receiving the dose of HepaGam B HBIG, blood glucose will be monitored in 3 manners. These will include two finger stick tests, one with a glucose-specific monitoring device and one with a glucose non-specific monitoring device; a venous blood glucose level; and a urine glucose test. Patients will receive the HBIG infusion and then immediately after the dose will have the same blood glucose tests repeated (finger sticks, venous glucose and urine glucose). Then at 60 minutes and 120 minutes after the dose is given, patients will again have finger stick tests with the glucose specific and glucose non-specific monitoring devices.
  HepaGam B (Hepatitis B Immune Globulin (HBIG)): Subjects will be gi
Arm/Group | Acute Phase | Chronic Phase
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No